CLINICAL TRIAL: NCT03744026
Title: A Study to Evaluate the Safety and the Efficacy of Transient Opening of the Blood-brain Barrier (BBB) by Low Intensity Pulsed Ultrasound With the SonoCloud-9 Implantable Device in Recurrent Glioblastoma Patients Eligible for Surgery and for Carboplatin Chemotherapy
Brief Title: Safety and Efficacy of Transient Opening of the Blood-brain Barrier (BBB) With the SonoCloud-9
Acronym: SC9-GBM-01
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: CarThera (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SC9-GBM-01
Record Dates: First submitted 2018-11-13; First posted 2018-11-16 (Actual); Last update posted 2022-09-07 (Actual); Status verified 2022-09

CONDITIONS: Glioblastoma, Adult
Keywords: Recurrent Glioblastoma; Carboplatin; Ultrasound; Blood-brain barrier; Glioblastoma; SonoCloud; Low Intensity Pulsed Ultrasound (LIPU)
MeSH Terms: conditions — Glioblastoma | interventions — Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- SonoCloud-9 Ultrasound + Carboplatin (Experimental): SonoCloud-9 Carboplatin: 6 cycles (every 4 weeks)
  Interventions: Device: SonoCloud-9; Drug: Carboplatin

INTERVENTIONS:
Device: SonoCloud-9 — Escalating numbers of ultrasound beams at constant acoustic pressure
Drug: Carboplatin — Dose of carboplatin infusion is AUC4-6

SUMMARY:
Recurrent glioblastoma (GBM) is a disease with high unmet clinical need. The standard of care for patients with GBM includes surgery, radiotherapy and chemotherapy. Despite this aggressive treatment, the overall median survival of patients with GBM remains at 15-20 months.

In more than 95% of cases, tumor recurrence is observed within 2 cm to 3 cm of the resection cavity within 4-7 months after initial treatments. One of the main causes of recurrence is the inability of chemotherapies to enter the brain from the systemic circulation due to the blood-brain barrier (BBB). The BBB is unique to cerebral blood vessels and blocks most drugs from entering the brain in sufficient concentrations.

The SonoCloud-9 (SC9) System delivers ultrasound to locally and transiently increase the permeability of the BBB to allow the passage of drugs into the cerebral parenchyma. The SC9 is dimensioned to cover the resection area and surrounding tissues in patients with recurrent GBM. The large sonicated volume covered by the SC9 device allows for broad BBB disruption and should allow for carboplatin chemotherapy to penetrate the surrounding tumor infiltrative area. By enhancing drug concentrations, it is hypothesized that further disease progression will be prevented.

DETAILED DESCRIPTION:
This will be an open-label, Phase 1/2a, multicenter, single-arm, interventional trial that will first evaluate the dose limiting toxicity (DLT) of escalating numbers of ultrasound beams at constant acoustic pressure using a standard escalation (Phase 1) and then confirm the safety and efficacy of BBB opening (Phase 2a expansion).

ELIGIBILITY:
Key Inclusion Criteria:

1. Age ≥ 18 years, able and willing to give signed and informed consent.
2. Patient with histologically proven recurrent de novo GBM:

   1. After at least a first-line standard of care (maximal safe resection, if feasible, radiation with temozolomide [TMZ], then TMZ);
   2. Any recurrence;
   3. Bevacizumab-naïve.*
3. Patient eligible for carboplatin-based chemotherapy.
4. Patient eligible for a surgical resection.
5. Maximal tumor diameter at inclusion (pre surgery) ≤ 70 mm in T1wMRI.
6. Patients should be stable, without evidence of a midline shift, significant peritumoral edema, or rapid progression of clinical symptoms.
7. Karnofsky performance status ≥ 70.
8. Patient receiving prednisone dose ≤ 40 mg (dexamethasone ≤ 6 mg) for at least 7 days.

Key Exclusion Criteria:

1. Multifocal tumor (unless all localized in a 70 mm diameter area).
2. Patients at risk of surgery site infection (2 or more previous craniotomies, neurosurgery within the last 3 months, poor skin condition, and/or previously infected surgical field).
3. Posterior fossa tumor.
4. Uncontrolled epilepsy.
5. Patients with evidence of uncontrolled intracranial pressure.
6. Patients with known intracranial aneurism or having presented intra-tumor spontaneous hemorrhage.
7. Patients with coils, clips, shunts, intravascular stents, and/or unremovable wafer, non resorbable dura substitute, or reservoirs.
8. Patients with medical need to continue antiplatelet therapy.
9. Patients with known or suspected active or chronic infections.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2019-02-18 (Actual); Primary Completion 2021-06-23 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLT) of number of activated ultrasound beams | 15 days after the first sonication treatment
  DLT will be evaluated using imaging (MRI) and clinical examination, as CTCAE that occurs within 2 weeks of the first sonication and that does not respond to optimal medical management (including steroids) within 7 days.
Blood-Brain Barrier (BBB) opening | At the end of the first three sonication treatments (treatment occurs every 4 weeks)
  BBB opening will be evaluated by contrast-enhanced T1w magnetic resonance imaging (MRI)

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed IDBAIH, MD, Principal Investigator — APHP
Locations (6):
- United States (2):
  - Northwestern University, Chicago, Illinois
  - MD Anderson Cancer Center, Houston, Texas
- France (4):
  - CHU, Angers
  - Hôpital Neurologique Pierre Wertheimer, Bron
  - Hôpital de La Timone, Marseille
  - Hôpital de la Pitié-Salpêtrière, Paris

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Carpentier A, Canney M, Vignot A, Reina V, Beccaria K, Horodyckid C, Karachi C, Leclercq D, Lafon C, Chapelon JY, Capelle L, Cornu P, Sanson M, Hoang-Xuan K, Delattre JY, Idbaih A. Clinical trial of blood-brain barrier disruption by pulsed ultrasound. Sci Transl Med. 2016 Jun 15;8(343):343re2. doi: 10.1126/scitranslmed.aaf6086. PMID 27306666
- [Derived] Sonabend AM, Gould A, Amidei C, Ward R, Schmidt KA, Zhang DY, Gomez C, Bebawy JF, Liu BP, Bouchoux G, Desseaux C, Helenowski IB, Lukas RV, Dixit K, Kumthekar P, Arrieta VA, Lesniak MS, Carpentier A, Zhang H, Muzzio M, Canney M, Stupp R. Repeated blood-brain barrier opening with an implantable ultrasound device for delivery of albumin-bound paclitaxel in patients with recurrent glioblastoma: a phase 1 trial. Lancet Oncol. 2023 May;24(5):509-522. doi: 10.1016/S1470-2045(23)00112-2. PMID 37142373
- See also: CarThera — http://www.carthera.eu